CLINICAL TRIAL: NCT00243971
Title: A Phase 3, Randomized, Open-Label, Two-Arm, Parallel-Group, Multicenter, Multinational Trial to Compare the Efficacy of Rotigotine Transdermal Patch to That of Ropinirole on Early Morning Motor Impairment and Sleep Disorders in Subjects With Early-Stage, Idiopathic Parkinson's Disease
Brief Title: A Trial to Compare the Efficacy of Rotigotine Transdermal Patch to That of Ropinirole on Early Morning Motor Impairment and Sleep Disorders in Subjects With Early-Stage, Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP0825; 2004-002609-66 (EudraCT Number)
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Parkinson's Disease
Keywords: EARLY-STAGE, IDIOPATHIC PARKINSON'S DISEASE
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Drug: SPM 962

SUMMARY:
The objective of this trial is to compare the effect of rotigotine (SPM 962) and ropinirole on the control of early morning motor impairment and sleep disorders in subjects with early-stage PD.

Subjects who meet eligibility criteria will be randomly assigned either to rotigotine transdermal patch or ropinirole tablets. Trial medication will be titrated for rotigotine and ropinirole until an individual optimal dose is achieved. Following a Titration period of up to 4 weeks in the rotigotine arm and 6 weeks in the ropinirole arm, subjects will be maintained on the optimal or maximal dose for 4 weeks. At the end of the Maintenance period, subjects will be given the opportunity to enter a 2-year rotigotine patch extension trial.

The first subject was enrolled in December 2004. The last subject was enrolled in June 2005. Last subject out is expected for October 2005. The trial is still ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Early-stage, idiopathic Parkinson's disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Monheim, Germany